CLINICAL TRIAL: NCT06881940
Title: Rationale and Design of a Cardiac Rehabilitation Program on the Prevention of Cardiotoxicity in Breast Cancer Patients Undergoing Treatment With Anthracyclines and/or Trastuzumab: A Randomized, Active Control Group, Open-Label Trial
Brief Title: Cardiac Rehabilitation Program on the Prevention of Cardiotoxicity in Breast Cancer Patients Undergoing Treatment With Anthracyclines and/or Trastuzumab
Acronym: CARPTOX-BC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Nilda Gladys Espinola Zavaleta, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-1488
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Cancer Therapy-Related Cardiac Dysfunction
Keywords: Rehabilitation; Breast Neoplasms; Cardiotoxicity; Trastuzumab; Anthracyclines
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Interventional Model: Active Control Group Interventional Model Description: The risk exposure factors for the experimental group and the control group are the same Masking: None (Open Label) Allocation: Randomized
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Participants randomized to observational arm will receive standard oncological follow up and care.
  Interventions: Other: No Rehabilitation Program
- Rehabilitation Program (Experimental): Intervention arm receives standard oncological follow up and care + Rehabilitation Program
  Interventions: Other: Rehabilitation Program

INTERVENTIONS:
Other: Rehabilitation Program — Three of the five weekly sessions will take place at the gym in the Functional Unit of Breast Tumors at INCAN, under the supervision of Physical and Sports Medicine specialists and three physical therapists. These sessions allow for personalized feedback, enabling participants to confidently perform prescribed aerobic exercises at home on the remaining two days.
  Each session starts with a 10- to 15-minute warm-up focused on joint mobility. Aerobic training is conducted at moderate intensity (40-59% VO2max or heart rate reserve), monitored with a Polar® FT1 device. Intensity is periodically adjusted based on the Borg Rating of Perceived Exertion and the talk test. Over 4-6 weeks, session duration will gradually increase to 90 minutes per week, remaining consistent thereafter.
  Following aerobic training, resistance exercises targeting major muscle groups are performed using gym machines and dumbbells. The program includes seven exercises, progressively increasing load over 3-4 weeks.
  Arms: Rehabilitation Program
Other: No Rehabilitation Program — The control group will continue standard oncological treatment in addition to general recommendations regarding diet and physical activity, but without a structured exercise protocol.
  Arms: Standard of care

SUMMARY:
This study aims to evaluate the effectiveness of a cardiac rehabilitation protocol, incorporating aerobic and resistance exercise, in reducing the incidence of cardiotoxicity in breast cancer patients receiving treatment with anthracyclines and/or trastuzumab through a randomized, active control group, open-label clinical trial.

DETAILED DESCRIPTION:
This is a randomized, open-label, with an active control group trial. This study adopts the main evaluation indicator being the incidence of cardiac dysfunction or heart failure as a manifestation of cardiovascular toxicity, assessed following the 2022 European Society of Cardiology (ESC) definitions for cancer-related therapy cardiac dysfunction (CTRCD).

Participants who pass the inclusion criteria through research will provide written informed consent to take part in the study. Once consent is obtained, participants will be randomly assigned to one of two study groups using a simple randomization process. This will be accomplished through a computer-generated random number sequence list, which will be managed by a designated investigator from the research team. The intervention group will receive standard oncological treatment combined with an aerobic and resistance exercise program, following the FITT principle (Frequency, Intensity, Type, and Time) for exercise prescription. Three out of five weekly sessions will be conducted per week. The control group will continue standard oncological treatment in addition to general recommendations regarding diet and physical activity but without a structured exercise protocol. During the treatment process, both branches of the trial will be followed over a 12 months period, with scheduled outpatient evaluations to assess biochemical parameters, a 12-lead electrocardiogram (ECG), a transthoracic echocardiogram (TTE), and a cardiopulmonary exercise test (CPET). Both the intervention and control groups will undergo these assessments at four key time points: baseline (defined as the time before the start of the chemotherapy regime and after the study enrollment), 3 months, 6 months, and 12 months post-initiation of chemotherapy. The main outcome of this clinical trial is a composite of incident cardiotoxicity, defined according to the ESC guidelines. Other cardiac function related indicators such as symptomatic congestive heart failure or asymptomatic but decreased left ventricular ejection fraction (LVEF) or global longitudinal strain (GLS) and changes in cardiac biomarkers will be evaluated to determine the occurrence of cardiac toxicity. Secondary outcomes assessed the impact on echocardiographic parameters of cardiac function, fluctuations in biomarkers and blood tests, cardiorespiratory performance, the impact of quality of life and explore the role of traditional cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 70 years will be considered eligible.
* Active residents of any municipality within Mexico City and the surrounding metropolitan area will qualify, conditioned that their maximum travel time from their residence to our recruitment center does not exceed three hours using private or public transportation. This criterion is established to ensure adherence to the protocol and availability for participation in the required interventions and assessments throughout the study.
* Patients diagnosed with early-stage or locally advanced breast cancer (stages I, II, or III, according to the TNM classification-Tumor, Node, Metastasis) who will undergo treatment with anthracyclines and/or adjuvant/neoadjuvant anti-HER2 therapy will be included. Participants must be scheduled to receive pharmacological treatment, ensuring that the study focuses on a population undergoing specific therapies for breast cancer management.
* Candidates must have the capacity, availability, and willingness to participate in an aerobic and resistance exercise program. Participants are required to possess both the physical ability and the willingness to actively engage in a structured exercise program, which includes aerobic and resistance activities essential to the study's objectives.
* Patients will provide informed written consent to participate in the study. To uphold ethical research principles and ensure the protection of participants' rights, all patients must voluntarily give their informed consent after receiving comprehensive information regarding the study's objectives, procedures, benefits, and potential risks.

Exclusion Criteria:

* Metastatic disease: Individuals with medical or imaging evidence of metastasis to any peripheral organ.
* Cardiovascular disease: Patients with a self-reported history of cardiovascular conditions, such as heart failure or uncontrolled hypertension, that may limit their ability to safely engage in physical activity. Additionally, those with peripheral arterial disease or valvular heart disease will not be eligible.
* Ischemic heart disease: Patients with a history of ischemic heart disease.
* Neurological disorders: Individuals with self-reported neurological diseases that significantly impair coordination, balance, or motor control, such as advanced Parkinson's disease, late-stage multiple sclerosis, or paralysis, making physical activity unsafe.
* Musculoskeletal conditions: Patients with self-reported musculoskeletal injuries or disorders that hinder physical activity, including fractures within the last five years, moderate to severe sprains, tendinitis, or severe arthritis.
* Uncontrolled systemic comorbidities: Individuals with decompensated systemic conditions, including heart failure, chronic kidney disease, or poorly controlled diabetes, will be excluded.
* Severe respiratory diseases: Patients with severe respiratory conditions that prevent physical exercise participation.
* Physical limitations: Individuals with mobility impairments or conditions requiring constant assistance for basic physical activities, such as those using assistive devices (e.g., wheelchairs, walkers) or with limb amputations, will not be eligible for participation.
* Severe psychiatric disorders: Patients with uncontrolled psychiatric conditions, including schizophrenia, severe bipolar disorder, or major depressive disorder, that may interfere with their ability to actively participate in a supervised exercise program.

Elimination Criteria:

* Voluntary withdrawal from the protocol.
* Development of severe cardiotoxicity requiring pharmacological treatment.
* Adverse reactions to chemotherapeutic agents.
* Disease progression according to the TNM classification during treatment.
* Failure to complete at least 80% of the prescribed adjuvant or neoadjuvant oncological treatment.
* Occurrence of adverse events during the study, such as falls or injuries.
* Death during the study period.
* Any accident related to the exercise protocol, including falls, sprains, or fractures.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiac dysfunction or heart failure as a manifestation of cardiovascular toxicity in the intervention group and control group | From 1 week before starting oncological treatment to 1 year after the start of the chemotherapy regimen
  Calculate the incidence of cardiotoxicity associated with anthracycline and/or trastuzumab treatment of two groups following the 2022 European Society of Cardiology (ESC) definitions for cancer-related therapy cardiac dysfunction (CTRCD). LVEF greater than 50% with a relative GLS decrease exceeding 15% and/or a new rise in cardiac biomarkers. LVEF will be determined using Simpson's biplane method, incorporating apical four- and two-chamber views, while 2D-GLS measurements will be performed via velocity vector imaging. All echocardiographic evaluations will be conducted using a Siemens-Acuson 2000 system by a single expert in echocardiography, with results subsequently verified by a second expert to ensure accuracy and reliability. The classification of symptomatic congestive heart failure encompasses, but is not limited to, the presence of one or more of the following clinical manifestations: moist crackles in the lungs, bilateral anterior tibial edema, or lip cyanosis.

SECONDARY OUTCOMES:
Impact on echocardiographic parameters | From 1 week before starting oncological treatment to 1 year after the start of the chemotherapy regimen
  This study aims to evaluate cardiac function by examining changes in echocardiographic parameters, including chamber volumes, diameters, diastolic function, right ventricular function, and both biventricular and auricular global longitudinal strain (GLS).
Modification in series of circulating cardiac biomarkers | From 1 week before starting oncological treatment to 1 year after the start of the chemotherapy regimen
  Classical biomarkers of cardiac injury: C-reactive protein, Troponin I, B-type natriuretic peptide (NT-Pro BNP).
Evaluation of cardiorespiratory performance | From 1 week before starting oncological treatment to 1 year after the start of the chemotherapy regimen
  The study will investigate modifications in cardiorespiratory fitness by measuring peak oxygen uptake (VO2max) through a cardiopulmonary exercise test (CPET) conducted on a bicycle ergometer with individualized workload adjustments.
Quality of Life Questionnaire: FACT-B | From 1 week before starting oncological treatment to 1 year after the start of the chemotherapy regimen
  Investigators should evaluate the quality of life of the patient with QOL questionnaire (FACT-B)
Explore the role of traditional cardiovascular risk factors | From 1 week before starting oncological treatment to 1 year after the start of the chemotherapy regimen
  This research will explore the role of conventional cardiovascular risk factors-including smoking, lipid levels, systemic arterial hypertension, diabetes, obesity, sedentary behavior, and the Framingham risk score-as potential mediators in the development of cardiotoxicity.

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cancerología (INCAN), Mexico City, Mexico City
  - National Institute of Cancerology (INCAN), Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: No
Can apply to researchers

REFERENCES:
- [Background] Kerrigan DJ, Reddy M, Walker EM, Cook B, McCord J, Loutfi R, Saval MA, Baxter J, Brawner CA, Keteyian SJ. Cardiac Rehabilitation Improves Fitness in Patients With Subclinical Markers of Cardiotoxicity While Receiving Chemotherapy: A RANDOMIZED CONTROLLED STUDY. J Cardiopulm Rehabil Prev. 2023 Mar 1;43(2):129-134. doi: 10.1097/HCR.0000000000000719. Epub 2022 Aug 4. PMID 35940850
- [Background] Viamonte SG, Joaquim AV, Alves AJ, Vilela E, Capela A, Ferreira C, Duarte BF, Rato ND, Teixeira MP, Tavares A, Santos M, Ribeiro F. Cardio-Oncology Rehabilitation for Cancer Survivors With High Cardiovascular Risk: A Randomized Clinical Trial. JAMA Cardiol. 2023 Dec 1;8(12):1119-1128. doi: 10.1001/jamacardio.2023.3558. PMID 37819656
- [Background] Diaz-Balboa E, Pena-Gil C, Rodriguez-Romero B, Cuesta-Vargas AI, Lado-Baleato O, Martinez-Monzonis A, Pedreira-Perez M, Palacios-Ozores P, Lopez-Lopez R, Gonzalez-Juanatey JR, Gonzalez-Salvado V. Exercise-based cardio-oncology rehabilitation for cardiotoxicity prevention during breast cancer chemotherapy: The ONCORE randomized controlled trial. Prog Cardiovasc Dis. 2024 Jul-Aug;85:74-81. doi: 10.1016/j.pcad.2024.02.002. Epub 2024 Feb 21. PMID 38395212
- [Background] Yang HL, Hsieh PL, Hung CH, Cheng HC, Chou WC, Chu PM, Chang YC, Tsai KL. Early Moderate Intensity Aerobic Exercise Intervention Prevents Doxorubicin-Caused Cardiac Dysfunction Through Inhibition of Cardiac Fibrosis and Inflammation. Cancers (Basel). 2020 Apr 28;12(5):1102. doi: 10.3390/cancers12051102. PMID 32354131
- [Background] Kouzi SA, Uddin MN. Aerobic Exercise Training as a Potential Cardioprotective Strategy to Attenuate Doxorubicin-Induced Cardiotoxicity. J Pharm Pharm Sci. 2016 Jul-Sep;19(3):399-410. doi: 10.18433/J3JS5R. PMID 27806245
- [Background] Yu AF, Jones LW. Breast cancer treatment-associated cardiovascular toxicity and effects of exercise countermeasures. Cardiooncology. 2016;2:1. doi: 10.1186/s40959-016-0011-5. Epub 2016 Feb 25. PMID 28133540
- [Background] Xie S, Sun Y, Zhao X, Xiao Y, Zhou F, Lin L, Wang W, Lin B, Wang Z, Fang Z, Wang L, Zhang Y. An update of the molecular mechanisms underlying anthracycline induced cardiotoxicity. Front Pharmacol. 2024 Jun 26;15:1406247. doi: 10.3389/fphar.2024.1406247. eCollection 2024. PMID 38989148
- [Background] Nebigil CG, Desaubry L. Updates in Anthracycline-Mediated Cardiotoxicity. Front Pharmacol. 2018 Nov 12;9:1262. doi: 10.3389/fphar.2018.01262. eCollection 2018. PMID 30483123
- [Background] Angsutararux P, Luanpitpong S, Issaragrisil S. Chemotherapy-Induced Cardiotoxicity: Overview of the Roles of Oxidative Stress. Oxid Med Cell Longev. 2015;2015:795602. doi: 10.1155/2015/795602. Epub 2015 Sep 29. PMID 26491536
- [Background] Herrmann J, Lenihan D, Armenian S, Barac A, Blaes A, Cardinale D, Carver J, Dent S, Ky B, Lyon AR, Lopez-Fernandez T, Fradley MG, Ganatra S, Curigliano G, Mitchell JD, Minotti G, Lang NN, Liu JE, Neilan TG, Nohria A, O'Quinn R, Pusic I, Porter C, Reynolds KL, Ruddy KJ, Thavendiranathan P, Valent P. Defining cardiovascular toxicities of cancer therapies: an International Cardio-Oncology Society (IC-OS) consensus statement. Eur Heart J. 2022 Jan 31;43(4):280-299. doi: 10.1093/eurheartj/ehab674. PMID 34904661
- [Background] Wang Y, Wang Y, Han X, Sun J, Li C, Adhikari BK, Zhang J, Miao X, Chen Z. Cardio-Oncology: A Myriad of Relationships Between Cardiovascular Disease and Cancer. Front Cardiovasc Med. 2022 Mar 17;9:727487. doi: 10.3389/fcvm.2022.727487. eCollection 2022. PMID 35369296
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Gilchrist SC, Barac A, Ades PA, Alfano CM, Franklin BA, Jones LW, La Gerche A, Ligibel JA, Lopez G, Madan K, Oeffinger KC, Salamone J, Scott JM, Squires RW, Thomas RJ, Treat-Jacobson DJ, Wright JS; American Heart Association Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Peripheral Vascular Disease. Cardio-Oncology Rehabilitation to Manage Cardiovascular Outcomes in Cancer Patients and Survivors: A Scientific Statement From the American Heart Association. Circulation. 2019 May 21;139(21):e997-e1012. doi: 10.1161/CIR.0000000000000679. PMID 30955352
- [Background] Lavin-Perez AM, Collado-Mateo D, Hinojo Gonzalez C, de Juan Ferre A, Ruisanchez Villar C, Mayo X, Jimenez A. High-intensity exercise prescription guided by heart rate variability in breast cancer patients: a study protocol for a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Mar 8;15(1):28. doi: 10.1186/s13102-023-00634-2. PMID 36890601
- [Background] Antunes P, Joaquim A, Sampaio F, Nunes C, Ascensao A, Vilela E, Teixeira M, Capela A, Amarelo A, Marques C, Viamonte S, Alves A, Esteves D. Effects of exercise training on cardiac toxicity markers in women with breast cancer undergoing chemotherapy with anthracyclines: a randomized controlled trial. Eur J Prev Cardiol. 2023 Jul 12;30(9):844-855. doi: 10.1093/eurjpc/zwad063. PMID 36857149
- [Background] Wilson RL, Christopher CN, Yang EH, Barac A, Adams SC, Scott JM, Dieli-Conwright CM. Incorporating Exercise Training into Cardio-Oncology Care: Current Evidence and Opportunities: JACC: CardioOncology State-of-the-Art Review. JACC CardioOncol. 2023 Oct 17;5(5):553-569. doi: 10.1016/j.jaccao.2023.08.008. eCollection 2023 Oct. PMID 37969654
- [Background] Wallace KB, Sardao VA, Oliveira PJ. Mitochondrial Determinants of Doxorubicin-Induced Cardiomyopathy. Circ Res. 2020 Mar 27;126(7):926-941. doi: 10.1161/CIRCRESAHA.119.314681. Epub 2020 Mar 26. PMID 32213135
- [Background] McGowan JV, Chung R, Maulik A, Piotrowska I, Walker JM, Yellon DM. Anthracycline Chemotherapy and Cardiotoxicity. Cardiovasc Drugs Ther. 2017 Feb;31(1):63-75. doi: 10.1007/s10557-016-6711-0. PMID 28185035
- [Background] Li H, Wang M, Huang Y. Anthracycline-induced cardiotoxicity: An overview from cellular structural perspective. Biomed Pharmacother. 2024 Oct;179:117312. doi: 10.1016/j.biopha.2024.117312. Epub 2024 Aug 20. PMID 39167843
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Background] Farmakis D. Is cardio-oncology a rapidly growing field of precision medicine? Eur J Heart Fail. 2020 Dec;22(12):2310-2313. doi: 10.1002/ejhf.2051. Epub 2020 Nov 24. No abstract available. PMID 33175447
- [Background] Dang CT, Yu AF, Jones LW, Liu J, Steingart RM, Argolo DF, Norton L, Hudis CA. Cardiac Surveillance Guidelines for Trastuzumab-Containing Therapy in Early-Stage Breast Cancer: Getting to the Heart of the Matter. J Clin Oncol. 2016 Apr 1;34(10):1030-3. doi: 10.1200/JCO.2015.64.5515. Epub 2016 Feb 1. No abstract available. PMID 26834055
- [Background] Denlinger CS, Sanft T, Baker KS, Broderick G, Demark-Wahnefried W, Friedman DL, Goldman M, Hudson M, Khakpour N, King A, Koura D, Lally RM, Langbaum TS, McDonough AL, Melisko M, Montoya JG, Mooney K, Moslehi JJ, O'Connor T, Overholser L, Paskett ED, Peppercorn J, Pirl W, Rodriguez MA, Ruddy KJ, Silverman P, Smith S, Syrjala KL, Tevaarwerk A, Urba SG, Wakabayashi MT, Zee P, McMillian NR, Freedman-Cass DA. Survivorship, Version 2.2018, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2018 Oct;16(10):1216-1247. doi: 10.6004/jnccn.2018.0078. PMID 30323092
- [Background] Camilli M, Cipolla CM, Dent S, Minotti G, Cardinale DM. Anthracycline Cardiotoxicity in Adult Cancer Patients: JACC: CardioOncology State-of-the-Art Review. JACC CardioOncol. 2024 Sep 17;6(5):655-677. doi: 10.1016/j.jaccao.2024.07.016. eCollection 2024 Oct. PMID 39479333